CLINICAL TRIAL: NCT00555711
Title: Monitoring Neural Tissues Properties by Modulated Imaging (MI)
Acronym: MI
Status: Withdrawn | Type: Observational
Why Stopped: no subject
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Mark Linskey, MD.,Department of Neurosurgery, University of California, Irvine
Other Study IDs: 20054775
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Brain Tumor
Keywords: Brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Modulated Imaging: Modulated Imaging
  Interventions: Device: Modulated Imaging

INTERVENTIONS:
Device: Modulated Imaging — Modulated Imaging

SUMMARY:
We have developed a safe, non-contact, intra-operative guidance system to optimize tumor resection in neurosurgery. The Modulated Imaging is non-contact optical imaging technology developed at the Beckman Laser Institute, UCI.

Compared to other imaging approaches, MI has the unique capability of performing both diffuse optical tomography and rapid, wide-field quantitative mapping of tissue optical properties within a single measurement platform.

Preliminary in vivo studies have shown that brain tumors, infiltrating tumor margins and normal brain may have intrinsically different optical properties.

DETAILED DESCRIPTION:
While compatible with time-modulation methods, MI alternatively uses spatially-modulated illumination for imaging of tissue constituents.

The Modulated Imaging system consists of

1. a light projection system that illuminates the tissue with spatial sinusoid patterns.
2. a CCD camera which collects the diffusely reflected light in a non-contact geometry. The wavelength of illumination can be selected by bandpass filtering of a broadband source,or by use of a monochromatic source.

Lastly, tissue fluorescence measurements can be performed by placing a combination of source-blocking and bandpass emission filters in front of the camera.

The diffusely reflected amplitude of the modulated wave carries both optical property (absorption, fluorescence, scattering) and depth information. Specifically, the sampling depth of the spatially-modulated wave is a function of the frequency of illumination and the tissue optical properties.

During neurosurgery when nervous tissue is exposed by the attending neurosurgeon, intraoperative pictures will be taken using the modulated imager by the investigators.

The imaging procedure may delay completion of the surgical case by an estimated 10 to 20 minutes. This is minimal prolongation considering most brain tumor resections take several hours.

The images acquired will be processed after the surgical procedure and will not be available to the surgeon during the operative procedure.

ELIGIBILITY:
Inclusion Criteria:

* All nervous system tumor patients who undergo a preoperative MRI,and undergoing central nervous system operative procedures for non tumor.

Exclusion Criteria:

* All emergency neurosurgical procedures.

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Brain Tissue Property | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Linskey, MD, Principal Investigator — University of California, Irvine; Bruce J Tromberg, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (2):
- United States (2):
  - Beckman Laser Institute,University of California,Irvine, Irvine, California
  - Neurosurgery department,University of California,Irvine, Orange, California